CLINICAL TRIAL: NCT02722993
Title: Efficacy of a Probiotic Product in Children With Antibiotic-associated Gastrointestinal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProGastro Kids 16
Record Dates: First submitted 2016-03-16; First posted 2016-03-30 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Antibiotic-associated Diarrhea
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Active Comparator)
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics
  Arms: Probiotics
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
To assess the effect of a probiotic product, when co-administered with antibiotics, on gastrointestinal symptoms following antibiotic treatment in children.

ELIGIBILITY:
Inclusion Criteria:

* Children at the age of 1-11 years that have been prescribed antibiotic treatment.
* Problems with loose stools during earlier antibiotic treatments.
* Children whose parents or legal caregivers have signed the informed consent to participate in the study.

Exclusion Criteria:

* Chronic intestinal disease, immunodeficiency or immunosuppressive treatment.
* Chronic or acute diarrheal disease.
* Use of laxatives the week before inclusion in the study.
* Antibiotic treatment for the last four weeks before inclusion in the study.
* Intake of probiotic products for the last two weeks before inclusion in the study.
* Known hypersensitivity to any of the ingredients in the probiotic product or the placebo (potato starch ± bacterial culture that may contain traces of soy).
* Patient requiring hospitalisation.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Number of loose/watery stools | 19-26 days

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Socha, Prof., Principal Investigator — Children's Memorial Health Institute, Warzaw, Poland
Locations (1):
- Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No